CLINICAL TRIAL: NCT05239286
Title: Comparison Between Conventional Fluid Management and Plethysmographic Variability Index Based Goal Directed Fluid Management in Patients Undergoing Spine Surgeries in Prone Position; A Randomized Control Trial.
Brief Title: Conventional Fluid Management vs Plethysmographic Variability Index -Based Goal Directed Fluid Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, Assisstant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-179-2020
Record Dates: First submitted 2022-01-21; First posted 2022-02-14 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Fluid Management During Elective Spine Surgeries
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group conventional (Active Comparator)
  Interventions: Procedure: General anaesthesia; Drug: Conventional fluid managment
- Group PVI (Experimental)
  Interventions: Procedure: General anaesthesia; Drug: PVI dependant goal directed fluid therapy

INTERVENTIONS:
Procedure: General anaesthesia — All patients in supine position will receive breathing 100% oxygen, induction of anaesthesia will be achieved using propofol (2 mg/Kg), 1-2 mcg/kg of fentanyl and atracurium (0.5 mg/Kg). Endotracheal tube will be inserted after 3 minutes of mask ventilation. Patients who will experience prolonged airway instrumentation due to a difficult intubation will be excluded from further data analysis because of excessive stimulation. Then mechanical ventilation will be performed using a tidal volume of 6-8 mL/kg of ideal body weight at an inspiratory to expiratory ratio of 1:2 without positive end-expiratory pressure. The ventilatory frequency will be adjusted to maintain an end-tidal carbon dioxide tension of 35-40 mmHg.
  Anaesthesia will be maintained by isoflurane (1-1.5%), atracurium 10 mg intravenous increments every 20 minutes and morphine 0.1 mg/kg intravenous will be given as a long acting analgesia.
Drug: Conventional fluid managment — Ringer solution at the dose of 5 ml/kg/h infused throughout the surgical procedure by taking the parameters such as Heart rate (HR), mean arterial pressure (MAP) and urine output, Hypotension was defined as a condition in which the MAP was below 30% of the baseline MAP of the patient. In this case, bolus of 250 ml crystalloids (0.9% NaCl) was given and in case of hypotension persistence, 5 mg I.V. ephedrine administered and repeated every 5 min till the MAP increased over 70% of baseline.
  Arms: Group conventional
Drug: PVI dependant goal directed fluid therapy — After the induction of anesthesia, Ringer solution infused at the dose of 2 ml/kg/h started as a basal rate of infusion. If the PVI was higher than 13% for more than 5 min, a 250-ml bolus of crystalloids administrated. If the PVI was still higher than 13% after the bolus, it was repeated every 5 min until the PVI was less than 13% and if MAP was below 30% of the baseline MAP of the patient 5 mg iv ephedrine was applied and repeated every 5 min to keep the MAP increased over 70% of baseline.
  In the cases where PVI was less than < 13% and if MAP was below 30% of the baseline MAP of the patient 5 mg iv ephedrine was applied and repeated every 5 min to keep the MAP increased over 70% of baseline.
  Then the patient was turned to prone position and the same steps according to Massimo readings were repeated.
  Arms: Group PVI

SUMMARY:
Plethysmographic variability index is a dynamic method for evaluation of volume status which depends on estimation of respiratory variations in pulse oximeter waveform amplitude. The PVI has been studied in various patient populations and clinical settings, and has been shown to reliably predict fluid responsiveness and guide fluid resuscitation.

conventional fluid management. Fluid replacement is managed according to clinical assessment, heart rate, arterial blood pressure and central venous pressure monitoring. However, clinical studies indicate that changes in ABP cannot be used for the monitoring of stroke volume and cardiac output. Another method is the goal-directed fluid management and it is based on individualized fluid management using static and dynamic parameters.

DETAILED DESCRIPTION:
This study aims to compare the conventional fluid managment and Plethysmographic Variability index based during elective spine surgeries in prone position.

the study hypothesize is: plethysmographic variability index (PVI) based fluid management is more accurate than conventional method in preventing hypovolemia ana hypotension associated with prone position.

The patients will be randomly assigned into two equal groups using computer-generated random numbers with closed envelop, each of which will include 33 patients.

Group conventional: (n=33) patients are in the conventional fluid management group.

Group PVI: (n=33) patients are in the PVI-based goal-directed fluid management group.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (18-65 years)

  * ASA I-II
  * Patients scheduled for elective lumbar spine surgeries (e.g.: Lumbar fixation and simple discectomy) under general anaesthesia in prone position.

Exclusion Criteria:

* • Operations which will last for less than 15 minutes. (e.g.: plate and screw adjustment or incomplete terminated surgery)

  * Patients with cardiac morbidities e.g. history of unstable angina, impaired contractility with ejection fraction < 40%, wall motional abnormalities or tight valvular lesions detected by echocardiography, previous cardiac operations or cardiac catherization with stent.
  * Patients with heart block and arrhythmia (atrial fibrillation and frequent ventricular or supraventricular premature beat).
  * Patient with decompensated respiratory disease (poor functional capacity, generalized wheezes, peripheral O2 saturation < 90% on room air).
  * Patients with peripheral vascular disease or long-standing DM affecting PVI readings.
  * Complicated surgeries (huge spine tumors, intraoperative vascular or neurological complications and prolonged durations more than 5 hours) or surgeries with massive blood loss (4 units of packed RBCs in 1 hour or replacement of 50% of total blood volume within 3 hours )
  * Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The total intraoperative crystalloid consumption | 3 hours
  the total volume of infused crystalloids intraoperatively.

SECONDARY OUTCOMES:
Plethysmographic variability index | 3 hours
  measured every 5 minutes intraoperatively taking in consideration these time points: in supine position in the operating room before induction of anaesthesia as a baseline reading (T0) -postinduction reading (T1) -after prone positioning(T2). Then every 30 minutes all through the operation.
perfusion index | 3 hours
  measured every 5 minutes intraoperatively taking in consideration these time points: in supine position in the operating room before induction of anaesthesia as a baseline reading (T0) -postinduction reading (T1) -after prone positioning(T2). Then every 30 minutes all through the operation.
mean arterial blood pressure | 3 hours
  measured every 5 minutes intraoperatively taking in consideration these time points: in supine position in the operating room before induction of anaesthesia as a baseline reading (T0) -postinduction reading (T1) -after prone positioning(T2). Then every 30 minutes all through the operation.
Heart rate | 3 hours
  measured every 5 minutes intraoperatively taking in consideration these time points: in supine position in the operating room before induction of anaesthesia as a baseline reading (T0) -postinduction reading (T1) -after prone positioning(T2). Then every 30 minutes all through the operation.
Blood lactate level | 3 hours
  It will be obtained after induction of anaesthesia (T1) and immediately postoperative in the recovery room (T2).
Total amount of intraoperative urine output | 3 hours
  • Oliguria (defined as a condition in which the intraoperative urine output < 0.5ml/kg/hr) will be recorded every hour and treated by boluses of 250 ml crystalloids (0.9% NaCl).
The need and the amount of intraoperative blood transfusion | 3 hours
  • The total amount of blood loss will be monitored and if exceed 20% of total blood volume blood transfusion will be started at a dose according to the estimated blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant M Abdelhamid, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Kasr Alaini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cesur S, Cardakozu T, Kus A, Turkyilmaz N, Yavuz O. Comparison of conventional fluid management with PVI-based goal-directed fluid management in elective colorectal surgery. J Clin Monit Comput. 2019 Apr;33(2):249-257. doi: 10.1007/s10877-018-0163-y. Epub 2018 Jun 14. PMID 29948666
- [Background] McDermid RC, Raghunathan K, Romanovsky A, Shaw AD, Bagshaw SM. Controversies in fluid therapy: Type, dose and toxicity. World J Crit Care Med. 2014 Feb 4;3(1):24-33. doi: 10.5492/wjccm.v3.i1.24. eCollection 2014 Feb 4. PMID 24834399
- [Background] Coutrot M, Joachim J, Depret F, Millasseau S, Nougue H, Mateo J, Mebazaa A, Gayat E, Vallee F. Noninvasive continuous detection of arterial hypotension during induction of anaesthesia using a photoplethysmographic signal: proof of concept. Br J Anaesth. 2019 May;122(5):605-612. doi: 10.1016/j.bja.2019.01.037. Epub 2019 Mar 11. PMID 30916032
- [Derived] Abdelhamid B, Matta M, Rady A, Adel G, Gamal M. Conventional fluid management versus plethysmographic variability index-based goal directed fluid management in patients undergoing spine surgery in the prone position - a randomised control trial. Anaesthesiol Intensive Ther. 2023;55(3):186-195. doi: 10.5114/ait.2023.130792. PMID 37728446